CLINICAL TRIAL: NCT00870675
Title: MRI of Ventriculomegaly: Morphology and Outcome
Brief Title: Magnetic Resonance Imaging (MRI) of Ventriculomegaly: Morphology and Outcome
Status: Completed | Type: Observational
Sponsor: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Collaborators: Beth Israel Deaconess Medical Center (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Deborah Levine, Professor of Radiology, National Institute for Biomedical Imaging and Bioengineering (NIBIB)
Other Study IDs: 2001-P-00842/6; NIH NIBIB 01998
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Ventriculomegaly
Keywords: Ventriculomegaly; ultrasound; MRI; fetus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ventriculomegaly: Pregnant women carrying a fetus with the ultrasound finding of enlarged ventricles (ventriculomegaly).

SUMMARY:
This study compares the accuracy of fast magnetic resonance imaging (MRI) using the half Fourier single shot rapid acceleration with relaxation enhancement technique to ultrasound in the diagnosis of fetal abnormalities. The investigators' specific aim is to perform MRI examinations with ultrafast MRI on fetuses with sonographic morphologic abnormalities. The investigators' hypotheses are that 1) MRI will demonstrate fetal morphologic abnormalities; and 2) MRI will add additional information to the sonographic diagnosis which may directly affect maternal and/or neonatal care.

DETAILED DESCRIPTION:
1. Study Design: This is a descriptive study looking at the potential for MRI to aid in the diagnosis of fetal ventriculomegaly. It will also compare the specificity of MRI and ultrasound in diagnosing additional morphologic abnormalities.

450 pregnant women in the second and third trimester with ventriculomegaly will be asked to participate. Sonograms will be performed according the American Institute of Ultrasound in Medicine/American College of Radiology guidelines. In addition, views will be obtained of the fetal face, lips, outflow tracts, hands, and feet.

The gestational age of the fetus, interpretation of the sonogram, with sonographic abnormality and specific diagnosis will be prospectively recorded. Other data collected will be age and ethnicity of the patient, results of chromosomal analysis during the current pregnancy, and gestational age at the time of original diagnosis of abnormality during this pregnancy.

After screening for contraindications to MRI examination patients will undergo a 20 minute MRI examination. MRI examinations will be performed with a 1.5 T superconductive system (SIEMENS VISION, Erlangen, Germany or General Electric Twin, Milwaukee) using a 4-8 element body phased-array coil and/or body coil. The minimum rise time will be 600 microseconds (for a 25 milliTesla preset gradient amplitude). The whole body specific absorption rate will be kept under 1.5 watt/kilogram. Patients will be positioned supine with their feet entering the magnet bore first to minimize feelings of claustrophobia. A scout view will be obtained, and fetal images will be obtained with half Fourier single shot fast spin echo imaging imaging in the fetal sagittal, coronal, and axial planes (echo spacing of 4.2 msec, echo time=60 msec, echo train length=72, 1 acquisition, 3-5 mm section thickness, 26 x 35 cm field of view, 128 x 256 acquisition matrix). The refocusing flip angle will be minimized to decrease the amount of radiofrequency power deposition. Fetal anomalies seen with MRI will be recorded prospectively with knowledge of the sonographic findings.

Interpretation of the sonograms will be performed independently of the MR results. Interpretation of MRI examinations will be performed by reviewers with knowledge of the results of the ultrasound. The principal investigator will then combine the results from the two modalities. When the diagnosis differs between the modalities, the images will be reviewed by three radiologists and a consensus will be reached. The results of the sonogram and MRI will be communicated to the referring physician. Affect of any change in patient care will be assessed.

Comparison of MR diagnoses will be made to sonographic diagnoses. Clinical and pathologic follow-up will be obtained postnatally on all fetuses enrolled in the study.

After the baby is born, at 3 months of age, the patients will be contacted by phone by one of the investigators at Beth Israel Deaconess Medical Center to see if they want to enroll their baby in the neonatal follow-up portion of the study. This involves cognitive and motor testing of the child at Boston's Children's Hospital at age 6 months, 1 year, 2 years and 3 years of age. If a head MR or head ultrasound has not been obtained for clinical indications, it will be offered to the patient at that time.

Timeline of postnatal follow-up Number of patient for postnatal follow-up at specified age* Patients Enrolled Peripartum follow-up 6 months 18 months 24 months 36 month Any age Year 1 90 68 18 18 Year 2 90 90 54 51 105 Year 3 90 90 54 51 49 154 Year 4 90 90 54 51 49 46 200 Year 5 90 90 54 51 49 46 200 Total 450 428 234 205 146 93 678

b. Data Analysis: This is primarily a descriptive study, comparing ultrasound and MR findings. Sonographic, MR, and postnatal diagnoses will be compared. Since this is a highly selected population, we cannot calculate sensitivity and specificity of each modality, but we can describe the type of findings visualized on one prenatal imaging modality that were not visualized on the other.

Data will be stored in an access database created specifically for this project

ELIGIBILITY:
Inclusion Criteria:

* Sonographic finding of ventriculomegaly
* Ability and willingness of the patient to provide informed consent and cooperate for the examination
* Absence of contraindications for MRI (claustrophobia, pacemaker, intracranial clips, intra-articular ocular debris)
* All patients must be greater than 18 years old and must be in the second or third trimester of pregnancy

Exclusion Criteria:

* Contraindications to MRI
* Age less than 18
* First trimester of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women carrying a fetus diagnosed by ultrasound as having ventriculomegaly.
Sampling Method: Non-Probability Sample
Enrollment: 434 (Actual)
Dates: Start 1996-01; Primary Completion 2009-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Live birth | within 6 months of enrollment
Postnatal imaging abnormalities | Within 3 years of birth
Postnatal developmental delay | Within 3 years of birth

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Levine, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Childrens Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Limperopoulos C, Robertson RL Jr, Khwaja OS, Robson CD, Estroff JA, Barnewolt C, Levine D, Morash D, Nemes L, Zaccagnini L, du Plessis AJ. How accurately does current fetal imaging identify posterior fossa anomalies? AJR Am J Roentgenol. 2008 Jun;190(6):1637-43. doi: 10.2214/AJR.07.3036. PMID 18492918
- [Result] Levine D, Feldman HA, Tannus JF, Estroff JA, Magnino M, Robson CD, Poussaint TY, Barnewolt CE, Mehta TS, Robertson RL. Frequency and cause of disagreements in diagnoses for fetuses referred for ventriculomegaly. Radiology. 2008 May;247(2):516-27. doi: 10.1148/radiol.2472071067. PMID 18430880
- [Result] Kazan-Tannus JF, Dialani V, Kataoka ML, Chiang G, Feldman HA, Brown JS, Levine D. MR volumetry of brain and CSF in fetuses referred for ventriculomegaly. AJR Am J Roentgenol. 2007 Jul;189(1):145-51. doi: 10.2214/AJR.07.2073. PMID 17579164
- [Result] Li Y, Estroff JA, Khwaja O, Mehta TS, Poussaint TY, Robson CD, Feldman HA, Ware J, Levine D. Callosal dysgenesis in fetuses with ventriculomegaly: levels of agreement between imaging modalities and postnatal outcome. Ultrasound Obstet Gynecol. 2012 Nov;40(5):522-9. doi: 10.1002/uog.11098. PMID 22262510
- [Result] Li Y, Estroff JA, Mehta TS, Robertson RL, Robson CD, Poussaint TY, Feldman HA, Ware J, Levine D. Ultrasound and MRI of fetuses with ventriculomegaly: can cortical development be used to predict postnatal outcome? AJR Am J Roentgenol. 2011 Jun;196(6):1457-67. doi: 10.2214/AJR.10.5422. PMID 21606314
- [Result] Pier DB, Levine D, Kataoka ML, Estroff JA, Werdich XQ, Ware J, Beeghly M, Poussaint TY, Duplessis A, Li Y, Feldman HA. Magnetic resonance volumetric assessments of brains in fetuses with ventriculomegaly correlated to outcomes. J Ultrasound Med. 2011 May;30(5):595-603. doi: 10.7863/jum.2011.30.5.595. PMID 21527607
- [Result] Li Y, Sansgiri RK, Estroff JA, Mehta TS, Poussaint TY, Robertson RL, Robson CD, Feldman HA, Barnewolt C, Levine D. Outcome of fetuses with cerebral ventriculomegaly and septum pellucidum leaflet abnormalities. AJR Am J Roentgenol. 2011 Jan;196(1):W83-92. doi: 10.2214/AJR.10.4434. PMID 21178039
- [Result] Senapati GM, Levine D, Smith C, Estroff JA, Barnewolt CE, Robertson RL, Poussaint TY, Mehta TS, Werdich XQ, Pier D, Feldman HA, Robson CD. Frequency and cause of disagreements in imaging diagnosis in children with ventriculomegaly diagnosed prenatally. Ultrasound Obstet Gynecol. 2010 Nov;36(5):582-95. doi: 10.1002/uog.7680. PMID 20499405
- [Result] Beeghly M, Ware J, Soul J, du Plessis A, Khwaja O, Senapati GM, Robson CD, Robertson RL, Poussaint TY, Barnewolt CE, Feldman HA, Estroff JA, Levine D. Neurodevelopmental outcome of fetuses referred for ventriculomegaly. Ultrasound Obstet Gynecol. 2010 Apr;35(4):405-16. doi: 10.1002/uog.7554. PMID 20069560